CLINICAL TRIAL: NCT04934683
Title: Tight Perioperative Blood Pressure Management to Reduce Serious Cardiovascular, Renal, and Cognitive Complications: The GUARDIAN Trial (Induction Agent Sub-Study Comparing Etomidate and Propofol)
Brief Title: The GUARDIAN Trial - Induction Agent Sub-Study
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Daniel Sessler, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: HSC-MS-24-1026 (induction)
Record Dates: First submitted 2021-06-15; First posted 2021-06-22 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-07

CONDITIONS: Major Surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Routine Blood Pressure Management and Etomidate Induction (Active Comparator): Etomidate will be used as the anesthetic induction agent.
  Interventions: Procedure: Routine Blood Pressure Management; Drug: Etomidate Induction
- Routine Blood Pressure Management and Propofol Induction (Active Comparator): Propofol will be used as the anesthetic induction agent.
  Interventions: Procedure: Routine Blood Pressure Management; Drug: Propofol Induction
- Tight Blood Pressure Management and Etomidate Induction (Active Comparator): Etomidate will be used as the anesthetic induction agent.
  Interventions: Procedure: Tight Blood Pressure Management; Drug: Etomidate Induction
- Tight Blood Pressure Management and Propofol Induction (Active Comparator): Propofol will be used as the anesthetic induction agent.
  Interventions: Procedure: Tight Blood Pressure Management; Drug: Propofol Induction

INTERVENTIONS:
Procedure: Routine Blood Pressure Management — Routine blood pressure control.
  Arms: Routine Blood Pressure Management and Etomidate Induction; Routine Blood Pressure Management and Propofol Induction
Procedure: Tight Blood Pressure Management — Tight blood pressure control.
  Arms: Tight Blood Pressure Management and Etomidate Induction; Tight Blood Pressure Management and Propofol Induction
Drug: Etomidate Induction — Anesthetic induction with etomidate.
  Arms: Routine Blood Pressure Management and Etomidate Induction; Tight Blood Pressure Management and Etomidate Induction
Drug: Propofol Induction — Anesthetic induction with propofol.
  Arms: Routine Blood Pressure Management and Propofol Induction; Tight Blood Pressure Management and Propofol Induction

SUMMARY:
This is a sub-study of the overall GUARDIAN trial (NCT04884802) in which some GUARDIAN trial participants will be additionally randomized to etomidate vs propofol for anesthetic induction.

DETAILED DESCRIPTION:
Participants in the underlying GUARDIAN trial (NCT04884802) will be randomized to: 1) routine intraoperative blood pressure management (routine pressure management); or 2) norepinephrine or phenylephrine infusion to maintain intraoperative MAP ≥85 mmHg (tight pressure management). Participants in this sub-study will be additionally randomized to etomidate or propofol for induction of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. At least 45 years old;
2. Scheduled for major noncardiac surgery expected to last at least 2 hours;
3. Having general anesthesia, neuraxial anesthesia, or the combination;
4. Expected to require at least overnight hospitalization (planned ICU admission is acceptable);
5. Are designated ASA physical status 2-4 (ranging from mild systemic disease through severe systemic disease that is a constant threat to life);
6. Expected to have direct intraoperative blood pressure monitoring with an arterial catheter;
7. Cared for by clinicians willing to follow the GUARDIAN protocol;
8. Subject to at least one of the following risk factors:

   1. Age >65 years;
   2. History of peripheral arterial disease;
   3. History of coronary artery disease;
   4. History of stroke or transient ischemic attack;
   5. Serum creatinine >175 μmol/L (>2.0 mg/dl) within 6 months;
   6. Diabetes requiring medication;
   7. Current smoking or 15 pack-year history of smoking tobacco;
   8. Scheduled for major vascular surgery;
   9. Body mass index ≥35 kg/m2;
   10. Preoperative high-sensitivity troponin T >14 ng/L or troponin I equivalent, defined as ≥15 ng/L (Abbott assay), 19 ng/L (Siemens assay, [Borges, unpublished]), or 25% of the 99% percentile for other assays - all within 6 months;
   11. B-type natriuretic protein (BNP) >80 ng/L or N-terminal B-type natriuretic protein (NTProBNP) >200 ng/L within six months.

Exclusion Criteria:

1. Are scheduled for carotid artery surgery;
2. Are scheduled for intracranial surgery;
3. Are scheduled for partial or complete nephrectomy;
4. Are scheduled for pheochromocytoma surgery;
5. Are scheduled for liver or kidney transplantation;
6. Require preoperative intravenous vasoactive medications;
7. Have a condition that precludes routine or tight blood pressure management such as surgeon request for relative hypotension;
8. Require beach-chair positioning;
9. Have a documented history of dementia;
10. Have language, vision, or hearing impairments that may compromise cognitive assessments;
11. Have contraindications to norepinephrine or phenylephrine per clinician judgement;
12. Have previously participated in the GUARDIAN trial.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6254 (Estimated)
Dates: Start 2021-07-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-04-25 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with a Composite of Major Perfusion-Related Complications | During the initial 30 days after major non-cardiac surgery
  The primary outcome is a composite of major perfusion-related complications (myocardial injury, stroke, non-fatal cardiac arrest, Stage 2-3 acute kidney injury, deep or organ-space infection, sepsis, and death) in the 30 days after major non-cardiac surgery.

SECONDARY OUTCOMES:
Number of Participants with Postoperative Delirium | During the initial 4 postoperative days
  The Postoperative Delirium Three-dimensional Confusion Assessment Method (3D CAM) will be used to assess for the presence of delirium over the initial four postoperative days.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I Sessler, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (11):
- United States (4):
  - University of Nebraska Medical Center, Omaha, Nebraska
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Main Campus, Cleveland, Ohio
- China (5):
  - Shanghai Ninth People's Hospital, Shanghai, Shanghai Municipality
  - Beijing Shijitan Hospital, Capital Medical University, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Shanghai Chest Hospital, Shanghai
  - West China Hospital, Sichuan
- University of Thessaly, Larissa, Greece
- National Defense College, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Each center will retain ownership of its own data. Publication of center-specific data will not be allowed until after the Main Trial Report is published, or two years have elapsed since enrollment of the last patient. The Executive Committee welcomes suggestions for sub-studies based on a partial or the full trial dataset. Sub-studies will be allocated based on importance and novelty of the proposals, and priority will be given to high-enrolling centers. However, all multi-center publications will be on a collaborative basis and include appropriate co-authors. The Executive Committee will do its best to be fair and equitable in assigning sub-studies.
  Data will be shared with external parties on a collaborative basis with approval of the Executive Committee and appropriate data-use agreements.